CLINICAL TRIAL: NCT04257253
Title: Effect of a Supervised Exercise Program on Paraspinal Muscle Morphology and Function in Patients With Chronic Low Back Pain: A Randomized Controlled Trial
Brief Title: Effect of a Supervised Exercise Program in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Concordia University, Montreal (Other)
Responsible Party: Principal Investigator, Maryse Fortin, Assistant Professor, Concordia University, Montreal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCER19-20-09
Record Dates: First submitted 2020-01-27; First posted 2020-02-05 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2023-03

CONDITIONS: Low Back Pain; Muscle Atrophy; Diagnostic Imaging; Exercise Therapy
Keywords: low back pain; paraspinal muscle; exercise; diagnostic imaging; randomized controlled trial
MeSH Terms: conditions — Low Back Pain; Muscular Atrophy; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Targeted exercise program (Experimental): Targeted motor control and isolated lumbar extensor strengthening exercises. Supervised 12-week program, 2 times a week.
  Interventions: Other: Targeted exercise program
- General exercise program (Active Comparator): General exercise program including upper body and lower body strengthening and flexibility exercises. Supervised 12-week program, 2 times a week.
  Interventions: Other: General exercise program

INTERVENTIONS:
Other: Targeted exercise program — Participants in this experimental intervention group will perform a combination of motor control and isolated lumbar extensor strenghtening exercises. The level of difficulty of the exercises will be progressed gradually. The intervention will last 12 weeks, and each participant will have 2 supervised exercise sessions per week.
  Arms: Targeted exercise program
Other: General exercise program — Participants in this active intervention group will perform a generalized exercise program comprising upper-body and lower-body and hip strengthening exercises, as well as flexibility. The level of difficulty of the exercises will be progressed gradually. The intervention will last 12 weeks, and each participant will have 2 supervised exercise sessions per week.
  Arms: General exercise program

SUMMARY:
This study evaluates the effect of a supervised exercise program on paraspinal muscle morphology and function, as well as disability/function in patients with non-specific chronic low back pain. Half of the participants will do a targeted paraspinal muscle exercise program, while the other half will do a general exercise program.

ELIGIBILITY:
Inclusion Criteria:

1. chronic nonspecific LBP (>3 months), defined as pain in the region between the lower ribs and gluteal folds, with or without leg pain
2. currently seeking care for LBP
3. between 18 and 60 years of age
4. English or French speaker
5. score of "moderate" or "severe" disability on the ODI questionnaire
6. do not currently engage in sports or fitness training specifically for the lower back muscles (3 months prior the beginning of the study).

Exclusion Criteria:

1. evidence of nerve root compression or reflex motor signs deficits (e.g. weakness, reflex changes, or sensory loss with same spinal nerve)
2. previous spinal surgery or vertebral fractures
3. other major lumbar spine structural abnormalities (e.g. spondylolysis, spondylolisthesis, or lumbar scoliosis >10°)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2022-01-11 (Actual)

PRIMARY OUTCOMES:
Change in multifidus muscle size (cross-sectional area) | Baseline, 6-week, 12-week
  Multifidus muscle cross-sectional area measurements will be obtained from magnetic resonance imaging (MRI) from L1 to L5 spinal levels.
Change in multifidus muscle fatty infiltration | Baseline, 6-week, 12-week
  Multifidus muscle fatty infiltration (composition) measurements will be obtained from magnetic resonance imaging (MRI) from L1 to L5 spinal levels.

SECONDARY OUTCOMES:
Change in12-item Short Form Health Survey (SF-12) | Baseline, 6-week, 12-week, 24-week
  The 12-item Short Form Health Survey (SF-12) is the condensed form of the previous 36-item Short Form Health Survey and is used to assess health-related quality of life.The 12-item survey consists of 8 domains that assess both physical and mental health composite scores (PCS and MCS). While the SF-12 is weighted and summed to provide an interpretable scale for both the PCS and MCS. The score of the 12 questions can range from 0 (worst level of health) to 100 (highest level of health).
Change in Oswestry Low Back Pain Disability Index (ODI) | Baseline, 6-week, 12-week, 24-week
  The ODI is used to measure the patient's level of disability in relation to LBP. It is a 10-item scale in which each item is rated from 0-6. Higher scores are indicative of greater disability.
Change in The International Physical Activity Questionnaire (IPAQ) | Baseline, 6-week, 12-week, 24-week
  The IPAQ is a self-reported log of metabolic equivalent (MET)-minutes per week. The level of physical activity is rated either vigorous, moderate, walking and sitting and must be assigned to the right category. The number of minutes per category is then added up and assessed.
Change in Tampa Scale of Kinesiophobia (TSK) | Baseline, 6-week, 12-week, 24-week
  The TSK measures pain-related fear in an individual through a 13-item scale. The scores range between 17 and 68 with increasing scores indicating a greater level of kinesiophobia.
Change in Visual Numerical pain rating scale (NPR) | Baseline, 6-week, 12-week, 24-week
  The NRP for pain is a rating system from 0 to 10 with 0 being no pain and 10 worst pain imaginable.
Change in The Pain Catastrophizing Scale (PCS) | Baseline, 6-week, 12-week, 24-week
  The PCS is a 13-item questionnaire that assesses the participant's level of catastrophizing. Each item is rated from 0-4 for a possible total of 52. The higher the score, the greater the level of catastrophizing.
Change in The Hospital Anxiety and Depression Scale (HADS) | Baseline, 6-week, 12-week, 24-week
  The HADS is a 14-item questionnaire used to assess a patient's level of depression and anxiety. Each item is rated from 0-3 with either depression or anxiety having scores between 0 and 21, with 21 being the highest level possible.
Change in Insomnia Severity Index (ISI) | Baseline, 6-week, 12-week, 24-week
  The ISI is a 7-item questionnaire used to assess sleep disturbances. Each item is rated from 0 to 4 and the total score is added. The higher the score, the greater the level of sleep disturbances.
Change in paraspinal muscle size (cross-sectional area) | Baseline, 6-week, 12-week
  Paraspinal muscle cross-sectional area measurements will be obtained from magnetic resonance imaging (MRI) from L1 to L5 spinal levels.
Change in paraspinal muscle fatty infiltration | Baseline, 6-week, 12-week
  Paraspinal muscle fatty infiltration (composition) measurements will be obtained from magnetic resonance imaging (MRI) from L1 to L5 spinal levels.
Change in multifidus muscle function (% thickness change) | Baseline, 6-week, 12-week
  Multifidus muscle function, expressed as the % thickness change from a rested to contracted position via contralateral arm lifts will be assessed by ultrasound.
Change in lumbar extensor muscle strength | Baseline, 6-week, 12-week
  lumbar extensor muscle strength will be assessed using a MedX Lumbar Isokinetic Dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- PERFORM Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No